CLINICAL TRIAL: NCT05445310
Title: Adjuvant Furmonertinib in Stage IA With High Risk Factors and Stage IB Non-small Cell Lung Cancer: a Prospective Single-arm Study
Brief Title: Adjuvant Furmonertinib in Stage IA With High Risk Factors and Stage IB Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AST-PMR2201
Record Dates: First submitted 2022-06-15; First posted 2022-07-06 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aflutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furmonertinib (Experimental): Patients will receive furmonertinib 80mg/d for 3 years or until disease recurrence or treatment cessation for other reasons.
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — Furmonertinib 80mg/d

SUMMARY:
This is a prospective, single arm study to investigate the efficacy and safety furmonertinib 80mg/d as adjuvant treatment for 3 years post surgery of stage IA with high-risk factors and stage IB non-small cell lung cancer. A total of 114 patients would be enrolled. The primary endpoint is the disease-free survival rate at 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Received radical resection of non-small cell lung cancer without prior anti-tumor therapies including radiotherapy, chemotherapy, target therapy and immunotherapy.
* Histologically diagnosed Non-small cell lung cancer based on the judgement of at least 2 pathologists.
* Stage IA with high risk factors including micropapillae or solid components, vascular invasion, spread through air spaces, low differentiation, tumor budding and insufficient lymph node dissection; Stage IB with or without high-risk factors. The pathological stage is based on the 8th edition of AJCC lung cancer staging.
* EGFR mutation positive according to NGS testing by tissue, including deletions in exon 19, L858R, S768I, G719X, L861Q, T790M mutations et al.
* ECOG performance status 0-1.
* Sufficient organ function in liver, renal, kidney and hematology.
* With written signed informed consent form, ability to report adverse events, and good adherence to clinical study.

Exclusion Criteria:

* Lung cancer with small cell or neuroendocrine cancer cell.
* EGFR exon 20 insertion positive.
* Concurrent with other diver mutations including alterations in ALK, ROS1, MET et al.
* Women who are pregnant or breastfeeding.
* Use of CYP3A4 strong depressant within 7 days or CYP3A4 strong inducer within 21 days prior to initial administration, use of other anti-tumor treatment including traditional Chinese medicine within 14 days before enrollment.
* Concurrent with other malignancies excluding carcinoma in situ.
* With uncontrolled systematic diseases such as active bleeding, unstable angina, heart infarction within 1 year, chronic heart failure and uncontrolled hypertension and diabetes mellitus; with active infection of HBV, HCV or HIV, or other infections requiring injection of antibiotics.
* Gastrointestinal disorders which may affect drug taking or absorption.
* With history of QT prolongation or relative risk factors including heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome et al.
* With history of interstitial lung disease or relative risk.
* Allergic to any component of furmonertinib tablet.
* Mental illness or drug abuse.
* Live vaccination within 30 days before enrollment.
* Other situation judged by investigator such as failure to follow the rules of study.
* Attending another study of investigational drug, or received other study drugs or medical devices with 4 weeks before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-08-06 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival rate at 3 years | 3 years following the first dose of study drug
  The rate of survival patients without disease recurrence at 3 years

SECONDARY OUTCOMES:
Overall survival rate at 3 years | 3 years following the first dose of study drug
  The rate of survival patients at 3 years
Median disease-free survival | Approximately 3 years following the first dose of study drugs
  The median time from the enrollment to the disease recurrence or death depending on the protocol
Median overall survival | Approximately 5 years following the first dose of study drugs
  The median time from the enrollment to death of any cause depending on the protocol
Adverse events | Approximately 3 years following the first dose of study drugs
  The number of patients with adverse events and the severity according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hopital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Blinded IPD are to be shared on the requirements of supervision department and overall results of the study are to be published on academic conferences and journals.